CLINICAL TRIAL: NCT00289484
Title: A Randomised, Double-Blind, Placebo Controlled Trial of Omega-3 Polyunsaturated Fatty Acid as an Augmentor of Antidepressant Medication for Major Depression.
Brief Title: A Study of Omega-3 as an Augmentor of Antidepressant Treatment for Major Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Your Health Inc. (Other); Sphere Healthcare (Industry); Ocean Nutrition (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05156
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Major Depression
Keywords: Mood disorder
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders | interventions — Docosahexaenoic Acids

INTERVENTIONS:
Drug: Omega-3 Polyunsaturated Fatty Acids

SUMMARY:
The purpose of this study is to determine whether augmentation of antidepressant medication with Omega-3 polyunsaturated fatty acids increases the speed and degree of improvement for patients with major depression

DETAILED DESCRIPTION:
The study will be a 4 week, parallel-group double blind randomised control trial of the efficacy pf Omega-3 as an augmentor of antidepressant treatment for depression. People aged between 18 and 65 with a first or new episode of depression warranting treatment with antidepressant medication will be recruited. In addition to their antidepressant medication, participants will be randomly allocated to receive either Omega-3 (fish oil) or placebo (paraffin oil)for 4 weeks. Participants will commence treatment with the antidepressant and Omega-3/placebo simultaneously. Participants will be followed up at 1,3 and 4 weeks and will be asked to rate their mood daily for the 4 week study period. Blood samples will be taken pre and post treatment to measure change in Omega-3 levels.

ELIGIBILITY:
Inclusion Criteria:

* Participants must present with a first or new episode of DSM IV non-psychotic major depression warranting treatment with antidepressant mediation.
* Must be able to give informed consent.

Exclusion Criteria:

* History of psychosis or mania/hypomania or personality disorder.
* Non-English speaking or otherwise unable to provide historical information.
* Having taken Omega-3 dietary supplements in the last 3 months.
* History of allergy to Omega-3 supplements, finfish or shellfish.
* Pregnancy, breast feeding or plans to become pregnant during course of study.
* Post-natal depression
* Current drug or alcohol abuse or dependence or history of abuse or dependence over the last 12 months.
* Unstable thyroid function
* Hepatic or renal impairment or other medical conditions that may interfere with the absorption and metabolism of Omega-3 polyunsaturated fatty acids
* Coagulopathy or anticoagulant treatment due to theoretical bleeding risk.
* Patients who, in the investigator's judgment pose a current serious suicidal or other safety risk, or patients who will not likely be able to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2006-02

PRIMARY OUTCOMES:
Change form pretreatment score on Depression Rating scale at 4 weeks

SECONDARY OUTCOMES:
Daily mood rating
Weekly measure of depression
Weekly measure of anxiety
Weekly measure of functional status

CONTACTS AND LOCATIONS:
Overall Officials: Gordon B Parker, Dsc MD PhD, Principal Investigator — Professor, School of Psychiatry UNSW and Exectutive Director, Black Dog Institute
Locations (1):
- The University of New South Wales/Black Dog Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Rees AM, Austin MP, Parker G. Role of omega-3 fatty acids as a treatment for depression in the perinatal period. Aust N Z J Psychiatry. 2005 Apr;39(4):274-80. doi: 10.1080/j.1440-1614.2005.01565.x. PMID 15777365
- [Background] Parker G, Gibson NA, Brotchie H, Heruc G, Rees AM, Hadzi-Pavlovic D. Omega-3 fatty acids and mood disorders. Am J Psychiatry. 2006 Jun;163(6):969-78. doi: 10.1176/ajp.2006.163.6.969. PMID 16741195
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au